CLINICAL TRIAL: NCT05230420
Title: Urine Bag Usage Versus Chest Drain Clamping After Lung Resection Surgeries
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Al-Quds University (Other)
Collaborators: Assiut University (Other); Tanta University (Other); European Institute of Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 02/REC-CT/2021
Record Dates: First submitted 2021-12-20; First posted 2022-02-08 (Actual); Last update posted 2022-02-08 (Actual); Status verified 2021-12

CONDITIONS: Pneumothorax and Air Leak; Pneumothorax; Pleura Injury; Pleural Effusion
MeSH Terms: conditions — Pneumothorax; Pleural Effusion | interventions — Constriction

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clamping (Experimental): This arm will undergo chest drain clamping after a certain criteria has been met. Four hours post clamping a chest x-ray will be made, and the presence of pneumothorax will be assessed. The chest drain will be removed only in the absence of pneumothorax, if pneumothorax persists patients will stay attached to the underwater seal
  Interventions: Other: Clamping
- Urine bag (Active Comparator): The second arm will be attached to a urine bag, and bag inflation will be measured after a certain criteria has been met. bag inflation will be assessed four hours after its attachment. Bag inflation indicates the persistence of an air leak, thus the absence of bag inflation indicates the removal of the chest drain
  Interventions: Other: Urine bag

INTERVENTIONS:
Other: Clamping — Clamping of chest tube
  Arms: Clamping
Other: Urine bag — Attachment of a urine bag to chest tube
  Arms: Urine bag

SUMMARY:
Investigators will compare two different approaches of postoperative drainage after the standard water-seal drain has been used efficiently; one is by using urine bag and check it get blown by the leaked air, two is by using clamping of the water seal drain. Investigators will compare them depending on several factors such as; cost effectiveness, hospital stay, duration of putting the drain and more, reinsertion of the chest tube and others.

ELIGIBILITY:
Inclusion Criteria:

* post lung resection patients (via Uniportal VATS only)
* Over the age of 18
* indicated chest tube

Exclusion Criteria:

* Under the age of 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-11-25 (Estimated); Study Completion 2022-12-25 (Estimated)

PRIMARY OUTCOMES:
Overall cost | 5 to 6 days
  The overall cost of the patient's hospital stay

SECONDARY OUTCOMES:
Number of participants with re-accumulation of air after chest tube clamping or attachment to the urine bag | up to 5 days
  An important side effect to be studied
total number of days with chest drain inserted | up to 5 days
  Number of days chest drain remained inserted
Number of chest x-rays | up to 5 days
  Total number of chest x-rays
Number of participants that faced other intervention associated side effects | up to 5 days
  Subcutaneous emphysema, tension pneumothorax and others
Number of participants with chest tube re-insertion | up to 5 days
  An important side effect

CONTACTS AND LOCATIONS:
Overall Officials: Firas Abuakar, MD, Principal Investigator — Thoracic Surgery Unit, Makassed Islamic Charitable Society Hospital, Jerusalem, Palestine; Osama Darras, MD candidate, Study Chair — Medical Research Club, faculty of medicine, Alquds University, Jerusalem, Palestine; Hadeel Abedalhameed, MD candidate, Study Chair — Medical Research Club, faculty of medicine, Alquds University, Jerusalem, Palestine; Rami Alaraj, MD candidate, Study Director — Medical Research Club, faculty of medicine, Alquds University, Jerusalem, Palestine; Rania Attiyeh, MD candidate, Study Chair — Medical Research Club, faculty of medicine, Alquds University, Jerusalem, Palestine
Locations (4):
- Egypt (2):
  - Assiut University, Asyut
  - Tanta University, Tanta
- European Institute of Oncology, Milan, Italy
- Makassed Hospital, East Jerusalem, Palestinian Territories

IPD SHARING:
Plan to Share IPD: No